CLINICAL TRIAL: NCT04933994
Title: Comparison of the Clinical and CT Features Between COVID-19 Pneumonia and H1N1 Influenza Pneumonia in Zhejiang, China
Brief Title: Comparison of COVID-19 and H1N1 Influenza Pneumonia
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Yueqing People's Hospital of Zhejiang Province (Unknown); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); Ruian People's Hospital of Zhejiang Province (Unknown); The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University (Unknown); First Affiliated Hospital of Zhejiang University (Other); Kecheng People's Hospital of Quzhou city, Zhejiang Province (Unknown); Pingyang People's Hospital of Zhejiang Province (Unknown); The First People's Hospital of Yuhang District, Hangzhou, Zhejiang Province (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-0187
Record Dates: First submitted 2021-06-17; First posted 2021-06-22 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2020-10

CONDITIONS: COVID-19; H1N1 Influenza
Keywords: COVID-19, H1N1, Tomography, X-ray computed
MeSH Terms: conditions — COVID-19; Orthomyxoviridae Infections | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Coronavirus disease; Influenza A(H1N1): two independent cohorts of COVID-19 pneumonia (n=405) and H1N1 influenza pneumonia (n=78) retrospectively, all patients were confirmed by RT-PCR. Four hundred and five cases of COVID-19 pneumonia were confirmed in nine hospitals of Zhejiang province, China from January 21 to February 20, 2020. Seventy-eight cases of H1N1 influenza pneumonia were confirmed in our hospital from January 1, 2017 to February 29, 2020.
  Interventions: Device: computed Tomography

INTERVENTIONS:
Device: computed Tomography — All cases were detected with computed Tomography

SUMMARY:
To explore the different clinical and CT features distinguishing COVID-19 from H1N1 influenza pneumonia.

DETAILED DESCRIPTION:
COVID-19 pneumonia patients showed less proportions of underlying diseases, fever and respiratory symptoms than those of H1N1 pneumonia patients (p<0.01). White blood cell count, neutrophilic granulocyte percentage, C-reactive protein, procalcitonin, D-Dimer and lactate dehydrogenase in H1N1 pneumonia patients were higher than those of COVID-19 pneumonia patients (p<0.05). H1N1 pneumonia were often symmetrically located in the dorsal part of lung inferior lobes, while COVID-19 pneumonia were unsually showed a peripheral but non-specific lobe distributions. Ground glass opacity was more common in COVID-19 pneumonia and consolidation lesions was more common in H1N1 pneumonia (p<0.01). COVID-19 pneumonia lesions showed a relative clear margin compared with H1N1 pneumonia. Crazy-paving pattern, thickening vessels, reversed halo sign and early fibrotic leisions were more common in COVID-19 pneumonia than H1N1 pneumonia (p<0.05). Pleural effusion in COVID-19 pneumonia was significantly less common than H1N1 pneumonia (p<0.01).

Compared with H1N1 pneumonia in Zhejiang, China, the clinical manifestations of COVID-19 pneumonia was more concealed with less underlying diseases and slighter respiratory symptoms. The more common CT manifestations of COVID-19 pneumonia included ground glass opacity with a relative clear margin, crazy-paving pattern, thickening vessels, reversed halo sign and early fibrotic leisions, while the less common CT manifestations of COVID-19 pneumonia included consolidation and pleural effusion.

ELIGIBILITY:
Inclusion Criteria:

* pneumonia

Exclusion Criteria:

* no pneumonia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pneumonia with COVID-19 pneumonia or H1N1 influenza
Sampling Method: Non-Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Comparison of the clinical and CT features between COVID-19 pneumonia and H1N1 influenza pneumonia in Zhejiang, China | 1 year
  one paper